CLINICAL TRIAL: NCT00257231
Title: Inflammation and the Host Response to Injury
Brief Title: Inflammation and the Host Response to Injury (Trauma)
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ronald G. Tompkins, Chief, Burns Service, Massachusetts General Hospital
Other Study IDs: 2 U54 GM062119_trauma; U54GM062119 (NIH)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Trauma; Burns; Multiple Organ Failure
Keywords: Immunity, innate; Inflammation; Genomics; Proteomics
MeSH Terms: conditions — Wounds and Injuries; Burns; Multiple Organ Failure; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, blood leukocyte nucleic acids (only RNA, no DNA)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to help improve our understanding of the biology involved in the body's response to serious trauma or burn injury. The host response to trauma and burns is a collection of physiological and pathophysiological processes that depend critically upon the regulation of the human innate immune system, with particular emphasis on the inflammatory component of that system. No single research center or small group of centers has the capacity to delineate the integrated response of this complex biological system, which involves multiple molecular and genetic interactions that vary in time. Our proposal promotes the identification of important dynamic relationships that regulate the integration of this complex biological system, with the expectation that this understanding will ultimately impact the diagnosis, prognosis, and treatment of the hospitalized, severely injured patient.

DETAILED DESCRIPTION:
This large-scale collaborative project provides the means to acquire the necessary new knowledge directly in humans. Knowledge will be acquired using diverse state-of-the-art genomic and proteomic technologies, a highly complex clinical, proteomic, and genomic database, as well as newly-developed, novel analytical tools to probe this complex dataset. Our analytical capabilities at the genomic and proteomic level are now rapidly evolving and our ability to link these genomic and proteomic data to pathways and functional modules will help us more closely link this cellular data to immunological processes and ultimately, to the phenotypic response (i.e., trajectory) in the injured host. As a result, potential interventions, whether through our Program or other funding mechanisms, can be more effectively designed.

ELIGIBILITY:
Inclusion criteria for enrollment in the trauma study are as follows:

* Blunt trauma without isolated head injury
* Absence of traumatic brain injury, defined as either AIS head <4 OR GCS motor >3 within 24 hours of injury
* Emergency Department arrival <=6 hours from time of injury
* Blood transfusion within 12 hours of injury
* Base deficit >=6 OR systolic blood pressure <90 mmHg within 60 minutes of emergency department arrival
* Fully or partially intact cervical spinal cord

All patients meeting these criteria are entered into the epidemiologic database and assessed for specific exclusion criteria to establish whether serial blood draws are warranted.

The presence of any of the following exclusion criteria disqualifies a subject from the trauma sampling study.

* Age < 16
* Anticipated survival of <24 hours from injury
* Anticipated survival <28 days due to pre-existing medical condition
* Inability to obtain first blood draw within first 12 hours after injury
* Traumatic brain injury; i.e., GCS ≤8 after ICU admission AND brain computerized tomography scan abnormality within 12 hours after injury
* Inability to obtain informed consent
* Pre-existing, ongoing immunosuppression - e.g. transplant recipient
* Pre-existing, ongoing immunosuppression - e.g. chronic high dose corticosteroids (>20 mg/prednisone-equivalents/day)
* Pre-existing, ongoing immunosuppression - e.g. oncolytic drug(s) therapy within the past 14 days
* Pre-existing, ongoing immunosuppression - e.g. HIV positive AND CD4 count <200 cells/mm3
* Possible requirement for early immunosuppression - e.g. significant likelihood of requiring high dose corticosteroids (e.g. spinal injury)
* Significant pre-existing organ dysfunction - lung: currently receiving home oxygen therapy, as documented in medical records
* Significant pre-existing organ dysfunction - heart: congestive heart failure, as documented in medical records
* Significant pre-existing organ dysfunction - renal: chronic renal failure (creatinine >2)
* Significant pre-existing organ dysfunction - liver: cirrhosis with portal hypertension or encephalopathy
* Patient injured while sampling enrollment temporarily on hold

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute hospitalized blunt trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 610 (Estimated)
Dates: Start 2003-11; Primary Completion 2013-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Time to death | Within 28 after trauma injury
Change in gene expression after trauma injury | Up to 28 days after trauma injury
Number and types of complications | Up to 28 days after trauma injury

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Tompkins, MD, ScD, Principal Investigator — Massachusetts General Hospital/Shriners Burn Hospital - Boston
Locations (4):
- United States (4):
  - Denver Health Medical Center at University of Colorado, Denver, Colorado
  - Presbyterian University Hospital at University of Pittsburgh, Pittsburgh, Pennsylvania
  - Southwestern Medical Center at University of Texas Southwestern, Dallas, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Curated and validated data are available to Consortium Members

REFERENCES:
- [Background] Siddiqui J, Remick DG. Improved sensitivity of colorimetric compared to chemiluminescence ELISAs for cytokine assays. J Immunoassay Immunochem. 2003;24(3):273-83. doi: 10.1081/IAS-120022937. PMID 12953972
- [Background] Shen Y, Jacobs JM, Camp DG 2nd, Fang R, Moore RJ, Smith RD, Xiao W, Davis RW, Tompkins RG. Ultra-high-efficiency strong cation exchange LC/RPLC/MS/MS for high dynamic range characterization of the human plasma proteome. Anal Chem. 2004 Feb 15;76(4):1134-44. doi: 10.1021/ac034869m. PMID 14961748
- [Background] Irimia D, Tompkins RG, Toner M. Single-cell chemical lysis in picoliter-scale closed volumes using a microfabricated device. Anal Chem. 2004 Oct 15;76(20):6137-43. doi: 10.1021/ac0497508. PMID 15481964
- [Background] Sethu P, Anahtar M, Moldawer LL, Tompkins RG, Toner M. Continuous flow microfluidic device for rapid erythrocyte lysis. Anal Chem. 2004 Nov 1;76(21):6247-53. doi: 10.1021/ac049429p. PMID 15516115
- [Background] Feezor RJ, Baker HV, Mindrinos M, Hayden D, Tannahill CL, Brownstein BH, Fay A, MacMillan S, Laramie J, Xiao W, Moldawer LL, Cobb JP, Laudanski K, Miller-Graziano CL, Maier RV, Schoenfeld D, Davis RW, Tompkins RG; Inflammation and Host Response to Injury, Large-Scale Collaborative Research Program. Whole blood and leukocyte RNA isolation for gene expression analyses. Physiol Genomics. 2004 Nov 17;19(3):247-54. doi: 10.1152/physiolgenomics.00020.2004. PMID 15548831
- [Background] Murthy SK, Sin A, Tompkins RG, Toner M. Effect of flow and surface conditions on human lymphocyte isolation using microfluidic chambers. Langmuir. 2004 Dec 21;20(26):11649-55. doi: 10.1021/la048047b. PMID 15595794
- [Background] Qian WJ, Jacobs JM, Camp DG 2nd, Monroe ME, Moore RJ, Gritsenko MA, Calvano SE, Lowry SF, Xiao W, Moldawer LL, Davis RW, Tompkins RG, Smith RD. Comparative proteome analyses of human plasma following in vivo lipopolysaccharide administration using multidimensional separations coupled with tandem mass spectrometry. Proteomics. 2005 Feb;5(2):572-84. doi: 10.1002/pmic.200400942. PMID 15627965
- [Background] Copeland S, Warren HS, Lowry SF, Calvano SE, Remick D; Inflammation and the Host Response to Injury Investigators. Acute inflammatory response to endotoxin in mice and humans. Clin Diagn Lab Immunol. 2005 Jan;12(1):60-7. doi: 10.1128/CDLI.12.1.60-67.2005. PMID 15642986
- [Background] Qian WJ, Monroe ME, Liu T, Jacobs JM, Anderson GA, Shen Y, Moore RJ, Anderson DJ, Zhang R, Calvano SE, Lowry SF, Xiao W, Moldawer LL, Davis RW, Tompkins RG, Camp DG 2nd, Smith RD; Inflammation and the Host Response to Injury Large Scale Collaborative Research Program. Quantitative proteome analysis of human plasma following in vivo lipopolysaccharide administration using 16O/18O labeling and the accurate mass and time tag approach. Mol Cell Proteomics. 2005 May;4(5):700-9. doi: 10.1074/mcp.M500045-MCP200. Epub 2005 Mar 7. PMID 15753121
- [Background] Cobb JP, Mindrinos MN, Miller-Graziano C, Calvano SE, Baker HV, Xiao W, Laudanski K, Brownstein BH, Elson CM, Hayden DL, Herndon DN, Lowry SF, Maier RV, Schoenfeld DA, Moldawer LL, Davis RW, Tompkins RG, Baker HV, Bankey P, Billiar T, Brownstein BH, Calvano SE, Camp D, Chaudry I, Cobb JP, Davis RW, Elson CM, Freeman B, Gamelli R, Gibran N, Harbrecht B, Hayden DL, Heagy W, Heimbach D, Herndon DN, Horton J, Hunt J, Laudanski K, Lederer J, Lowry SF, Maier RV, Mannick J, McKinley B, Miller-Graziano C, Mindrinos MN, Minei J, Moldawer LL, Moore E, Moore F, Munford R, Nathens A, O'keefe G, Purdue G, Rahme L, Remick D, Sailors M, Schoenfeld DA, Shapiro M, Silver G, Smith R, Stephanopoulos G, Stormo G, Tompkins RG, Toner M, Warren S, West M, Wolfe S, Xiao W, Young V; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. Application of genome-wide expression analysis to human health and disease. Proc Natl Acad Sci U S A. 2005 Mar 29;102(13):4801-6. doi: 10.1073/pnas.0409768102. Epub 2005 Mar 21. PMID 15781863
- [Background] Toner M, Irimia D. Blood-on-a-chip. Annu Rev Biomed Eng. 2005;7:77-103. doi: 10.1146/annurev.bioeng.7.011205.135108. PMID 16004567
- [Background] Calvano SE, Xiao W, Richards DR, Felciano RM, Baker HV, Cho RJ, Chen RO, Brownstein BH, Cobb JP, Tschoeke SK, Miller-Graziano C, Moldawer LL, Mindrinos MN, Davis RW, Tompkins RG, Lowry SF; Inflamm and Host Response to Injury Large Scale Collab. Res. Program. A network-based analysis of systemic inflammation in humans. Nature. 2005 Oct 13;437(7061):1032-7. doi: 10.1038/nature03985. Epub 2005 Aug 31. PMID 16136080
- [Background] Storey JD, Xiao W, Leek JT, Tompkins RG, Davis RW. Significance analysis of time course microarray experiments. Proc Natl Acad Sci U S A. 2005 Sep 6;102(36):12837-42. doi: 10.1073/pnas.0504609102. Epub 2005 Sep 2. PMID 16141318
- [Background] Shen Y, Kim J, Strittmatter EF, Jacobs JM, Camp DG 2nd, Fang R, Tolie N, Moore RJ, Smith RD. Characterization of the human blood plasma proteome. Proteomics. 2005 Oct;5(15):4034-45. doi: 10.1002/pmic.200401246. PMID 16152657
- [Background] De AK, Miller-Graziano CL, Calvano SE, Laudanski K, Lowry SF, Moldawer LL, Remick DG Jr, Rajicic N, Schoenfeld D, Tompkins RG. Selective activation of peripheral blood T cell subsets by endotoxin infusion in healthy human subjects corresponds to differential chemokine activation. J Immunol. 2005 Nov 1;175(9):6155-62. doi: 10.4049/jimmunol.175.9.6155. PMID 16237112
- [Background] Nathens AB, Johnson JL, Minei JP, Moore EE, Shapiro M, Bankey P, Freeman B, Harbrecht BG, Lowry SF, McKinley B, Moore F, West M, Maier RV; Inflammation and the Host Response to Injury Investigators. Inflammation and the Host Response to Injury, a large-scale collaborative project: Patient-Oriented Research Core--standard operating procedures for clinical care. I. Guidelines for mechanical ventilation of the trauma patient. J Trauma. 2005 Sep;59(3):764-9. No abstract available. PMID 16361929
- [Background] Brownstein BH, Logvinenko T, Lederer JA, Cobb JP, Hubbard WJ, Chaudry IH, Remick DG, Baker HV, Xiao W, Mannick JA. Commonality and differences in leukocyte gene expression patterns among three models of inflammation and injury. Physiol Genomics. 2006 Feb 14;24(3):298-309. doi: 10.1152/physiolgenomics.00213.2005. Epub 2005 Dec 20. PMID 16478828
- [Background] Liu T, Qian WJ, Gritsenko MA, Xiao W, Moldawer LL, Kaushal A, Monroe ME, Varnum SM, Moore RJ, Purvine SO, Maier RV, Davis RW, Tompkins RG, Camp DG 2nd, Smith RD; Inflammation and the Host Response to Injury Large Scale Collaborative Research Programm. High dynamic range characterization of the trauma patient plasma proteome. Mol Cell Proteomics. 2006 Oct;5(10):1899-913. doi: 10.1074/mcp.M600068-MCP200. Epub 2006 May 9. PMID 16684767
- [Background] Minei JP, Nathens AB, West M, Harbrecht BG, Moore EE, Shapiro MB, Bankey PE, Johnson JL, Freeman B, McKinley BA, Moore FA, Maier RV; Inflammation and the Host Response to Injury Large Scale Collaborative Research Program Investigators. Inflammation and the Host Response to Injury, a Large-Scale Collaborative Project: patient-oriented research core--standard operating procedures for clinical care. II. Guidelines for prevention, diagnosis and treatment of ventilator-associated pneumonia (VAP) in the trauma patient. J Trauma. 2006 May;60(5):1106-13; discussion 1113. doi: 10.1097/01.ta.0000220424.34835.f1. No abstract available. PMID 16688078
- [Background] Moore FA, McKinley BA, Moore EE, Nathens AB, West M, Shapiro MB, Bankey P, Freeman B, Harbrecht BG, Johnson JL, Minei JP, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Inflammation and the Host Response to Injury, a large-scale collaborative project: patient-oriented research core--standard operating procedures for clinical care. III. Guidelines for shock resuscitation. J Trauma. 2006 Jul;61(1):82-9. doi: 10.1097/01.ta.0000225933.08478.65. No abstract available. PMID 16832253
- [Background] Sethu P, Moldawer LL, Mindrinos MN, Scumpia PO, Tannahill CL, Wilhelmy J, Efron PA, Brownstein BH, Tompkins RG, Toner M. Microfluidic isolation of leukocytes from whole blood for phenotype and gene expression analysis. Anal Chem. 2006 Aug 1;78(15):5453-61. doi: 10.1021/ac060140c. PMID 16878882
- [Background] Qian WJ, Jacobs JM, Liu T, Camp DG 2nd, Smith RD. Advances and challenges in liquid chromatography-mass spectrometry-based proteomics profiling for clinical applications. Mol Cell Proteomics. 2006 Oct;5(10):1727-44. doi: 10.1074/mcp.M600162-MCP200. Epub 2006 Aug 3. PMID 16887931
- [Background] West MA, Shapiro MB, Nathens AB, Johnson JL, Moore EE, Minei JP, Bankey PE, Freeman B, Harbrecht BG, McKinley BA, Moore FA, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Inflammation and the host response to injury, a large-scale collaborative project: Patient-oriented research core-standard operating procedures for clinical care. IV. Guidelines for transfusion in the trauma patient. J Trauma. 2006 Aug;61(2):436-9. doi: 10.1097/01.ta.0000232517.83039.c4. No abstract available. PMID 16917462
- [Background] Rajicic N, Finkelstein DM, Schoenfeld DA; Inflammation Host Response to Injury Research Program Investigators. Survival analysis of longitudinal microarrays. Bioinformatics. 2006 Nov 1;22(21):2643-9. doi: 10.1093/bioinformatics/btl450. Epub 2006 Oct 10. PMID 17032680
- [Background] Laudanski K, Miller-Graziano C, Xiao W, Mindrinos MN, Richards DR, De A, Moldawer LL, Maier RV, Bankey P, Baker HV, Brownstein BH, Cobb JP, Calvano SE, Davis RW, Tompkins RG. Cell-specific expression and pathway analyses reveal alterations in trauma-related human T cell and monocyte pathways. Proc Natl Acad Sci U S A. 2006 Oct 17;103(42):15564-9. doi: 10.1073/pnas.0607028103. Epub 2006 Oct 10. PMID 17032758
- [Background] Nathens AB, McMurray MK, Cuschieri J, Durr EA, Moore EE, Bankey PE, Freeman B, Harbrecht BG, Johnson JL, Minei JP, McKinley BA, Moore FA, Shapiro MB, West MA, Tompkins RG, Maier RV. The practice of venous thromboembolism prophylaxis in the major trauma patient. J Trauma. 2007 Mar;62(3):557-62; discussion 562-3. doi: 10.1097/TA.0b013e318031b5f5. PMID 17414328
- [Background] Leek JT, Storey JD. Capturing heterogeneity in gene expression studies by surrogate variable analysis. PLoS Genet. 2007 Sep;3(9):1724-35. doi: 10.1371/journal.pgen.0030161. Epub 2007 Aug 1. PMID 17907809
- [Background] Lederer JA, Brownstein BH, Lopez MC, Macmillan S, Delisle AJ, Macconmara MP, Choudhry MA, Xiao W, Lekousi S, Cobb JP, Baker HV, Mannick JA, Chaudry IH; Inflammation and the Host Response to Injury Collaborative Research Program Participants. Comparison of longitudinal leukocyte gene expression after burn injury or trauma-hemorrhage in mice. Physiol Genomics. 2008 Feb 19;32(3):299-310. doi: 10.1152/physiolgenomics.00086.2007. Epub 2007 Nov 6. PMID 17986522
- [Background] Harbrecht BG, Minei JP, Shapiro MB, Nathens AB, Moore EE, West MA, Bankey PE, Cuschieri J, Johnson JL, Maier RV; Inflammation and the Host Response to Injury Scale Collaborative Research Project. Inflammation and the host response to injury, a large-scale collaborative project: patient-oriented research core-standard operating procedures for clinical care: VI. Blood glucose control in the critically ill trauma patient. J Trauma. 2007 Sep;63(3):703-8. doi: 10.1097/TA.0b013e31811eadea. No abstract available. PMID 18073622
- [Background] Shapiro MB, West MA, Nathens AB, Harbrecht BG, Moore FA, Bankey PE, Freeman B, Johnson JL, McKinley BA, Minei JP, Moore EE, Maier RV; Inflammation and the Host Response to Injury Large Scale Collaborative Research Project. V. Guidelines for sedation and analgesia during mechanical ventilation general overview. J Trauma. 2007 Oct;63(4):945-50. doi: 10.1097/TA.0b013e318142d21b. No abstract available. PMID 18090028
- [Background] Polpitiya AD, Qian WJ, Jaitly N, Petyuk VA, Adkins JN, Camp DG 2nd, Anderson GA, Smith RD. DAnTE: a statistical tool for quantitative analysis of -omics data. Bioinformatics. 2008 Jul 1;24(13):1556-8. doi: 10.1093/bioinformatics/btn217. Epub 2008 May 3. PMID 18453552
- [Background] Cuschieri J, Freeman B, O'Keefe G, Harbrecht BG, Bankey P, Johnson JL, Minei JP, Sperry J, West M, Nathens A, Moore EE, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Inflammation and the host response to injury a large-scale collaborative project: patient-oriented research core standard operating procedure for clinical care X. Guidelines for venous thromboembolism prophylaxis in the trauma patient. J Trauma. 2008 Oct;65(4):944-50. doi: 10.1097/TA.0b013e3181826df7. No abstract available. PMID 18849816
- [Background] O'Keefe GE, Shelton M, Cuschieri J, Moore EE, Lowry SF, Harbrecht BG, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Inflammation and the host response to injury, a large-scale collaborative project: patient-oriented research core--standard operating procedures for clinical care VIII--Nutritional support of the trauma patient. J Trauma. 2008 Dec;65(6):1520-8. doi: 10.1097/TA.0b013e3181904b0c. No abstract available. PMID 19077652
- [Background] West MA, Moore EE, Shapiro MB, Nathens AB, Cuschieri J, Johnson JL, Harbrecht BG, Minei JP, Bankey PE, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. Inflammation and the host response to injury, a large-scale collaborative project: patient-oriented research core--standard operating procedures for clinical care VII--Guidelines for antibiotic administration in severely injured patients. J Trauma. 2008 Dec;65(6):1511-9. doi: 10.1097/TA.0b013e318184ee35. PMID 19077651
- [Background] Evans HL, Cuschieri J, Moore EE, Shapiro MB, Nathens AB, Johnson JL, Harbrecht BG, Minei JP, Bankey PE, Maier RV, West MA; Inflammation and Host Response to Injury Investigators. Inflammation and the host response to injury, a Large-Scale Collaborative Project: patient-oriented research core standard operating procedures for clinical care IX. Definitions for complications of clinical care of critically injured patients. J Trauma. 2009 Aug;67(2):384-8. doi: 10.1097/TA.0b013e3181ad66a7. No abstract available. PMID 19667895
- [Background] Warren HS, Tompkins RG, Moldawer LL, Seok J, Xu W, Mindrinos MN, Maier RV, Xiao W, Davis RW. Mice are not men. Proc Natl Acad Sci U S A. 2015 Jan 27;112(4):E345. doi: 10.1073/pnas.1414857111. Epub 2014 Dec 24. No abstract available. PMID 25540422
- [Result] Escobar GA, Cheng AM, Moore EE, Johnson JL, Tannahill C, Baker HV, Moldawer LL, Banerjee A. Stored packed red blood cell transfusion up-regulates inflammatory gene expression in circulating leukocytes. Ann Surg. 2007 Jul;246(1):129-34. doi: 10.1097/01.sla.0000264507.79859.f9. PMID 17592301
- [Result] Russom A, Sethu P, Irimia D, Mindrinos MN, Calvano SE, Garcia I, Finnerty C, Tannahill C, Abouhamze A, Wilhelmy J, Lopez MC, Baker HV, Herndon DN, Lowry SF, Maier RV, Davis RW, Moldawer LL, Tompkins RG, Toner M; Inflammation and Host Response to Injury Large Scale Collaborative Research Program. Microfluidic leukocyte isolation for gene expression analysis in critically ill hospitalized patients. Clin Chem. 2008 May;54(5):891-900. doi: 10.1373/clinchem.2007.099150. Epub 2008 Mar 28. PMID 18375483
- [Result] Sperry JL, Frankel HL, Nathens AB, O'keefe GE, Cuschieri J, Moore EE, Maier RV, Minei JP; Inflammation and the Host Response to Injury Investigators. Characterization of persistent hyperglycemia: what does it mean postinjury? J Trauma. 2009 Apr;66(4):1076-82. doi: 10.1097/TA.0b013e31817db0de. PMID 19359917
- [Result] Hayden D, Lazar P, Schoenfeld D; Inflammation and the Host Response to Injury Investigators. Assessing statistical significance in microarray experiments using the distance between microarrays. PLoS One. 2009 Jun 16;4(6):e5838. doi: 10.1371/journal.pone.0005838. PMID 19529777
- [Result] Warren HS, Elson CM, Hayden DL, Schoenfeld DA, Cobb JP, Maier RV, Moldawer LL, Moore EE, Harbrecht BG, Pelak K, Cuschieri J, Herndon DN, Jeschke MG, Finnerty CC, Brownstein BH, Hennessy L, Mason PH, Tompkins RG; Inflammation and Host Response to Injury Large Scale Collaborative Research Program. A genomic score prognostic of outcome in trauma patients. Mol Med. 2009 Jul-Aug;15(7-8):220-7. doi: 10.2119/molmed.2009.00027. Epub 2009 Apr 10. PMID 19593405
- [Result] Rajicic N, Finkelstein DM, Schoenfeld DA; Inflammation and Host Response to Injury Research Program Investigators. Analysis of the relationship between longitudinal gene expressions and ordered categorical event data. Stat Med. 2009 Sep 30;28(22):2817-32. doi: 10.1002/sim.3665. PMID 19618375
- [Result] Cobb JP, Moore EE, Hayden DL, Minei JP, Cuschieri J, Yang J, Li Q, Lin N, Brownstein BH, Hennessy L, Mason PH, Schierding WS, Dixon DJ, Tompkins RG, Warren HS, Schoenfeld DA, Maier RV. Validation of the riboleukogram to detect ventilator-associated pneumonia after severe injury. Ann Surg. 2009 Oct;250(4):531-9. doi: 10.1097/SLA.0b013e3181b8fbd5. PMID 19730236
- [Result] Neal MD, Cushieri J, Rosengart MR, Alarcon LH, Moore EE, Maier RV, Minei JP, Billiar TR, Peitzman AB, Sperry JL; Inflammation and Host Response to Injury Investigators. Preinjury statin use is associated with a higher risk of multiple organ failure after injury: a propensity score adjusted analysis. J Trauma. 2009 Sep;67(3):476-82; discussion 482-4. doi: 10.1097/TA.0b013e3181ad66bb. PMID 19741387
- [Result] Irimia D, Mindrinos M, Russom A, Xiao W, Wilhelmy J, Wang S, Heath JD, Kurn N, Tompkins RG, Davis RW, Toner M. Genome-wide transcriptome analysis of 150 cell samples. Integr Biol (Camb). 2009 Jan;1(1):99-107. doi: 10.1039/b814329c. Epub 2008 Nov 12. PMID 20023796
- [Result] Kotz KT, Xiao W, Miller-Graziano C, Qian WJ, Russom A, Warner EA, Moldawer LL, De A, Bankey PE, Petritis BO, Camp DG 2nd, Rosenbach AE, Goverman J, Fagan SP, Brownstein BH, Irimia D, Xu W, Wilhelmy J, Mindrinos MN, Smith RD, Davis RW, Tompkins RG, Toner M; Inflammation and the Host Response to Injury Collaborative Research Program. Clinical microfluidics for neutrophil genomics and proteomics. Nat Med. 2010 Sep;16(9):1042-7. doi: 10.1038/nm.2205. Epub 2010 Aug 29. PMID 20802500
- [Result] Xu W, Seok J, Mindrinos MN, Schweitzer AC, Jiang H, Wilhelmy J, Clark TA, Kapur K, Xing Y, Faham M, Storey JD, Moldawer LL, Maier RV, Tompkins RG, Wong WH, Davis RW, Xiao W; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. Human transcriptome array for high-throughput clinical studies. Proc Natl Acad Sci U S A. 2011 Mar 1;108(9):3707-12. doi: 10.1073/pnas.1019753108. Epub 2011 Feb 11. PMID 21317363
- [Result] Minei JP, Cuschieri J, Sperry J, Moore EE, West MA, Harbrecht BG, O'Keefe GE, Cohen MJ, Moldawer LL, Tompkins RG, Maier RV; Inflammation and the Host Response to Injury Collaborative Research Program. The changing pattern and implications of multiple organ failure after blunt injury with hemorrhagic shock. Crit Care Med. 2012 Apr;40(4):1129-35. doi: 10.1097/CCM.0b013e3182376e9f. PMID 22020243
- [Result] Xiao W, Mindrinos MN, Seok J, Cuschieri J, Cuenca AG, Gao H, Hayden DL, Hennessy L, Moore EE, Minei JP, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Brownstein BH, Mason PH, Baker HV, Finnerty CC, Jeschke MG, Lopez MC, Klein MB, Gamelli RL, Gibran NS, Arnoldo B, Xu W, Zhang Y, Calvano SE, McDonald-Smith GP, Schoenfeld DA, Storey JD, Cobb JP, Warren HS, Moldawer LL, Herndon DN, Lowry SF, Maier RV, Davis RW, Tompkins RG; Inflammation and Host Response to Injury Large-Scale Collaborative Research Program. A genomic storm in critically injured humans. J Exp Med. 2011 Dec 19;208(13):2581-90. doi: 10.1084/jem.20111354. Epub 2011 Nov 21. PMID 22110166
- [Result] Cuschieri J, Johnson JL, Sperry J, West MA, Moore EE, Minei JP, Bankey PE, Nathens AB, Cuenca AG, Efron PA, Hennessy L, Xiao W, Mindrinos MN, McDonald-Smith GP, Mason PH, Billiar TR, Schoenfeld DA, Warren HS, Cobb JP, Moldawer LL, Davis RW, Maier RV, Tompkins RG; Inflammation and Host Response to Injury, Large Scale Collaborative Research Program. Benchmarking outcomes in the critically injured trauma patient and the effect of implementing standard operating procedures. Ann Surg. 2012 May;255(5):993-9. doi: 10.1097/SLA.0b013e31824f1ebc. PMID 22470077
- [Result] Desai KH, Tan CS, Leek JT, Maier RV, Tompkins RG, Storey JD; Inflammation and the Host Response to Injury Large-Scale Collaborative Research Program. Dissecting inflammatory complications in critically injured patients by within-patient gene expression changes: a longitudinal clinical genomics study. PLoS Med. 2011 Sep;8(9):e1001093. doi: 10.1371/journal.pmed.1001093. Epub 2011 Sep 13. PMID 21931541
- [Result] Warner EA, Kotz KT, Ungaro RF, Abouhamze AS, Lopez MC, Cuenca AG, Kelly-Scumpia KM, Moreno C, O'Malley KA, Lanz JD, Baker HV, Martin LC, Toner M, Tompkins RG, Efron PA, Moldawer LL. Microfluidics-based capture of human neutrophils for expression analysis in blood and bronchoalveolar lavage. Lab Invest. 2011 Dec;91(12):1787-95. doi: 10.1038/labinvest.2011.94. Epub 2011 Sep 19. PMID 21931299
- [Result] Seok J, Warren HS, Cuenca AG, Mindrinos MN, Baker HV, Xu W, Richards DR, McDonald-Smith GP, Gao H, Hennessy L, Finnerty CC, Lopez CM, Honari S, Moore EE, Minei JP, Cuschieri J, Bankey PE, Johnson JL, Sperry J, Nathens AB, Billiar TR, West MA, Jeschke MG, Klein MB, Gamelli RL, Gibran NS, Brownstein BH, Miller-Graziano C, Calvano SE, Mason PH, Cobb JP, Rahme LG, Lowry SF, Maier RV, Moldawer LL, Herndon DN, Davis RW, Xiao W, Tompkins RG; Inflammation and Host Response to Injury, Large Scale Collaborative Research Program. Genomic responses in mouse models poorly mimic human inflammatory diseases. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):3507-12. doi: 10.1073/pnas.1222878110. Epub 2013 Feb 11. PMID 23401516
- [Result] Zhou JY, Krovvidi RK, Gao Y, Gao H, Petritis BO, De AK, Miller-Graziano CL, Bankey PE, Petyuk VA, Nicora CD, Clauss TR, Moore RJ, Shi T, Brown JN, Kaushal A, Xiao W, Davis RW, Maier RV, Tompkins RG, Qian WJ, Camp DG 2nd, Smith RD; Inflammation and the Host Response to Injury Large Scale Collaborative Research Program. Trauma-associated human neutrophil alterations revealed by comparative proteomics profiling. Proteomics Clin Appl. 2013 Aug;7(7-8):571-83. doi: 10.1002/prca.201200109. Epub 2013 May 22. PMID 23589343
- [Result] Cuenca AG, Gentile LF, Lopez MC, Ungaro R, Liu H, Xiao W, Seok J, Mindrinos MN, Ang D, Baslanti TO, Bihorac A, Efron PA, Cuschieri J, Warren HS, Tompkins RG, Maier RV, Baker HV, Moldawer LL; Inflammation and Host Response to Injury Collaborative Research Program. Development of a genomic metric that can be rapidly used to predict clinical outcome in severely injured trauma patients. Crit Care Med. 2013 May;41(5):1175-85. doi: 10.1097/CCM.0b013e318277131c. PMID 23388514
- [Result] Warren HS, Tompkins RG, Mindrinos MN, Xiao W, Davis RW. Reply to Cauwels et al.: Of men, not mice, and inflammation. Proc Natl Acad Sci U S A. 2013 Aug 20;110(34):E3151. doi: 10.1073/pnas.1308943110. No abstract available. PMID 24137663
- [Result] Tompkins RG, Warren HS, Mindrinos MN, Xiao W, Davis RW. Reply to Osterburg et al.: To study human inflammatory diseases in humans. Proc Natl Acad Sci U S A. 2013 Sep 3;110(36):E3371. doi: 10.1073/pnas.1307452110. No abstract available. PMID 24137798
- See also: Information about the study and its goals. Contains links to study related publications, resources, and participating institutions — http://www.gluegrant.org